CLINICAL TRIAL: NCT06318689
Title: In Situ Exploration of Vascular Function in Vasoplegic Shock Following Cardiac Surgery With Cardiopulmonary Bypass
Acronym: Vaso-shock
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0211/OB
Record Dates: First submitted 2024-02-23; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Surgical Procedures
Keywords: Cardiopulmonary Bypass; Vasoplegia; Glycocalyx; Vascular function
MeSH Terms: conditions — Vasoplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Blood samples will be collected using 1 tube of 5 mL EDTA at inclusion and at 48 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess in situ vascular function, glycocalyx and microcirculation in postoperative vasoplegic shock following cardiac surgery with cardiopulmonary bypass.

The main question is to investigate the relationship between NO-dependent vasomotor reserve and the presence of vasoplegic shock following cardiac surgery with cardiopulmonary bypass.

Participants will have two visits, during which a number of non-invasive examinations will be carried out to study glycocalyx, microcirculation and vascular function. Biological and morphological data will be collected up to 3 months after inclusion, as well as information on treatments administered and outcome.

Researchers will compare a group of patients with vasoplegic shock against a group without vasoplegic shock in order to study possible alterations in function in the vasoplegic shock group.

DETAILED DESCRIPTION:
Objective : the primary objective of this study is to explore in situ the glycocalyx, the microcirculation and vascular function in postoperative vasoplegic shock following cardiac surgery with CPB. Secondary objectives are to study links between vascular function and damage to the glycocalyx and microcirculation and patient prognosis, in particular their impact on fluid balance.

Method :

Constitution of a single-centre prospective cohort study of 124 patients. Patients hospitalised in the cardiac intensive care unit after cardiac surgery with CPB will be consecutively included from 4 to 24 hours after surgery: 62 patients with vasoplegic shock (noradrenaline > 0.05µg/kg/min for at least 4 hours and after correction of any hypovolaemia), 62 patients without vasoplegic shock.

Endothelial function will be assessed using the flow-mediated dilation (FMD) method to test brachial artery vasodilation mediated by nitric oxide (NO) after induced ischemia. Microcirculation and glycocalyx will be evaluated using GlycoCheck, providing several measurements of microcirculation and glycocalyx using Sidestream Dark Field technology (mucosal illumination by a green LED and continuous x20 magnification video recording at the sublingual mucosa level). Various endothelial and inflammatory markers will also be measured (VCAM-1, syndecan, endothelin, interleukin-6).

Each patient will be assessed at inclusion and 48 hours using GlycoCheck, FMD, and endothelial measurements, then followed through their medical records for 90 days, where a follow-up call will be conducted to assess outcomes. Collected information will include routine care data (morphological data, vital signs, laboratory tests, fluid balance, scores, treatments, surgical data).

Both groups will be compared using statistical tests, and risk factors for developing vasoplegic shock will be explored through logistic regression. Univariable analysis followed by multivariable logistic regression with backward data inclusion will then be performed to identify risk factors for vasoplegic syndrome within the entire cohort (necessarily including FMD and GlycoCheck). A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years old
* Patient undergoing cardiac surgery with cardiopulmonary bypass
* Hospitalised in a cardiac surgical unit, between 4 and 24 hours after the end of cardiopulmonary bypass, after volemic optimisation

Exclusion Criteria:

* Sepsis at inclusion
* Cardiac transplant
* Circulatory assistance
* Known alteration of the microcirculation
* Any condition contraindicating measurement via Glycocheck or flux mediated dilatation measurement
* New surgery within 48 hours of the operation
* Person deprived of liberty by an administrative or judicial decision or person placed under legal protection / sub-guardianship or guardianship
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 80 years old hospitalised in the cardiac intensive care unit after cardiac surgery requiring cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Association between the percentage of brachial artery variation measured by the flow-mediated vasodilation method and the presence of vasoplegic shock at incusion. | At inclusion
  Association between the percentage of brachial artery variation measured by the flow-mediated vasodilation method and the presence of vasoplegic shock.

SECONDARY OUTCOMES:
Association between the percentage of brachial artery variation measured by the flow-mediated vasodilation method and the presence of vasoplegic shock at 48 hours. | At 48 hours
  Association between the percentage of brachial artery variation measured by the flow-mediated vasodilation method and the presence of vasoplegic shock.
Pefused boundary region (PBR, µm) obtained from Glycocheck with the presence of vasoplegic shock. | At inclusion and at 48 hours
  Pefused boundary region is an index given by the Glycocheck, a reflection of the alteration of the glycocalyx.
  The higher the value, the more impaired the glycocayx.
Microvascular blood flow (10^3 microns^3 / sec / mm^2) obtained from Glycocheck with the presence of vasoplegic shock | At inclusion and at 48 hours
  Microvascular blood flow (10^3 microns^3 / sec / mm^2), given by the Glycocheck, is an estimation of the microcirculation. The lower the value, the more it indicates a deterioration in microcirculation.
Total density (number of 10 micron long vessel segments with diameter of 4 to 25 microns per tissue surface area /mm^2) obtained from Glycocheck with the presence of vasoplegic shock | At inclusion and at 48 hours
  Total density (number of 10 micron long vessel segments with diameter of 4 to 25 microns per tissue surface area /mm^2), given by the Glycocheck, is an estimation of the density ot the vessels. The lower the value, the more it indicates a deterioration in microcirculation.
Endothelial function markers (Endothelin-1, pg/mL) with the presence of vasoplegic shock | At inclusion and at 48 hours
  Endothelin-1 (pg/ml), indicates vasoconstriction, will be measured by ELISA.
Endothelial function markers (syndecan-1, pg/mL) with the presence of vasoplegic shock | At inclusion and at 48 hours
  Endothelin-1 (pg/ml), indicates endothelium ateration, will be measured by ELISA.
Endothelial function markers (interleukin-6, pg/mL) with the presence of vasoplegic shock | At inclusion and at 48 hours
  Interleukin-6 (pg/ml), indicates inflammation, will be measured by ELISA.
Endothelial function markers (VCAM-1, pg/mL) with the presence of vasoplegic shock | At inclusion and at 48 hours
  VCAM-1 (pg/ml), indicates endothelium ateration, will be measured by ELISA.
Multivariate analysis explaining the occurrence of vasoplegic shock. | At inclusion and at 48 hours
  Model constructed from variables found to be associated in univariate analysis.
Multivariate analysis explaining the occurrence of an altered perfused boundary region (µm). | At inclusion and at 48 hours
  Model constructed from variables found to be associated in univariate analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel EB BESNIER, PHD, Principal Investigator — CHU Rouen
Locations (1):
- Rouen University Hospital, Rouen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided